CLINICAL TRIAL: NCT02897492
Title: Rapid and Highly Sensitive Detection of Fluorescently-labeled Troponin in Patients Admitted With Chest Pain
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, rambam75, Dr Shadi Hamoud, Rambam Health Care Campus
Other Study IDs: Rapid troponin detection
Record Dates: First submitted 2016-08-29; First posted 2016-09-13 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood testing in a newly described method — To exploit detection strategy termed "Magnetic Modulation Biosensing", or MMB) to develop a novel, low-cost platform that can detect biomarkers, such as proteins and specific DNA sequences, rapidly and directly from real samples at very low concentrations.

SUMMARY:
Patients with chest pain may have postponed or missed diagnosis of acute coronary events due to relatively late detection of troponin elevation. The study will investigate a new diagnostic method for early detection of even minimal troponin elevation in patients admitted with chest pain.

DETAILED DESCRIPTION:
Patients with chest pain may have postponed or missed diagnosis of acute coronary events due to relatively late detection of troponin elevation. The study will investigate a new diagnostic method for early detection of even minimal troponin elevation in patients admitted with chest pain.

A new diagnostic method will be applicated in the recent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years old or older
2. Admitted to Rambam health campus for the investigation of chest pain

Exclusion Criteria:

1. No exclusion criteria will be applied

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects will be patients admitted to Rambam health campus for the investigation of chest pain. Five m"l blood will be collected for troponin assay. No further intervention will be applied for subjects. Blood will be centrifuged and plasma separated for study purposes (detailed in "methods"- section 3.2.1.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Time to detect troponin elevation | sixty to 120 minutes

IPD SHARING:
Plan to Share IPD: Yes